CLINICAL TRIAL: NCT05936970
Title: Prospective, Multi-Center, Observational, Whole Blood Specimen Collection Study in Participants with Rheumatoid Arthritis with Inadequate Response or Intolerance to a DMARD Starting a New BDMARD or TsDMARD Treatment +/- CsDMARD
Status: Recruiting | Type: Observational
Sponsor: Aqtual, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PRIMA - 102
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood & processed plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults diagnosed with RA: Adults diagnosed with RA who are planning to initiate a new bDMARD +/- csDMARD or tsDMARD +/- csDMARD treatment

SUMMARY:
The primary goal of this study is to assess a cfDNA-based blood test using genetic, transcriptomic and/or epigenetic information to help doctors predict the best treatment options for rheumatoid arthritis (RA) patients with inadequate response or intolerance to previous therapies.

DETAILED DESCRIPTION:
PRIMA - 102 aims to predict response to bDMARD or tsDMARD therapy through analysis of cfDNA in blood. PRIMA - 102 will enroll participants with inadequate response or intolerance to previous therapies. Participants will undergo screening and baseline visits, followed by the initiation of new bDMARD or tsDMARD therapy per standard of care. The study will evaluate treatment response and disease activity at a 12-week follow-up visit. Blood will be drawn and Clinical Outcome Assessments performed at baseline and at the 12-week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and provide written informed consent.
* Male or female ≥18 years of age at enrollment.
* Diagnosis of Rheumatoid Arthritis at the time of enrollment.
* Prior treatment with at least 1 csDMARD, bDMARD, or tsDMARD
* Planning to initiate a new bDMARD (+/- csDMARD) or tsDMARD (+/- csDMARD), within 1 month after enrollment.
* Moderate to high Clinical Disease Activity Index (CDAI) of (>10) with a minimum 4 tender joints and 4 swollen joints at the time of screening.

Exclusion Criteria:

* Unsuitable for participation in the opinion of the principal investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with RA who are planning to initiate a new bDMARD +/- csDMARD or tsDMARD +/- csDMARD treatment
Sampling Method: Probability Sample
Enrollment: 1410 (Estimated)
Dates: Start 2023-06-29 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Response Prediction | Approximately 3 months
  This study aims to identify cfDNA signatures that predict response to specific bDMARD or tsDMARD therapies for RA treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Abdueva, Study Director — CEO
Locations (1):
- Arthritis and Osteoporosis Consultants of the Carolinas, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided